CLINICAL TRIAL: NCT01693315
Title: A Phase 2a, Randomized, Double-masked, Placebo-controlled, Dose-escalation Study of AMA0076 in Topical Ocular Formulation for Safety, Tolerability and Efficacy in Reduction of Intraocular Pressure in Subjects With Ocular Hypertension or Primary Open-angle Glaucoma
Brief Title: Multiple Dose-escalation Study of AMA0076 in Patients With Ocular Hypertension or Primary Open-angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amakem, NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMA0076-201
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Glaucoma; Ocular Hypertension; Eye Disease
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 - AMA0076 Dose A (or vehicle) (Experimental): Consecutive, eligible subjects who meet the inclusion/exclusion criteria in each cohort will be randomized to active or placebo (vehicle) in a 4:1 allocation ratio (12 active : 3 placebo).
  Interventions: Drug: AMA0076; Drug: Placebo
- Cohort 2: AMA0076 Dose B (or vehicle) (Experimental): Consecutive, eligible subjects who meet the inclusion/exclusion criteria in each cohort will be randomized to active or placebo (vehicle) in a 4:1 allocation ratio (12 active : 3 placebo).
  Interventions: Drug: AMA0076; Drug: Placebo
- Cohort 3: AMA0076 Dose C (or vehicle) (Experimental): Consecutive, eligible subjects who meet the inclusion/exclusion criteria in each cohort will be randomized to active or placebo (vehicle) in a 4:1 allocation ratio (20 active : 5 placebo).
  Interventions: Drug: AMA0076; Drug: Placebo
- Cohort 4: AMA0076 Dose D (or vehicle) (Experimental): Consecutive, eligible subjects who meet the inclusion/exclusion criteria in each cohort will be randomized to active or placebo (vehicle) in a 4:1 allocation ratio (20 active : 5 placebo).
  Interventions: Drug: AMA0076; Drug: Placebo

INTERVENTIONS:
Drug: AMA0076
Drug: Placebo

SUMMARY:
The objective of this dose-escalation study is to evaluate the safety, tolerability and efficacy of AMA0076 in reduction of intraocular pressure in subjects with ocular hypertension or primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria include:

1. Adults 30-85 years of age
2. Diagnosis of either ocular hypertension or primary open-angle glaucoma in both eyes
3. Not receiving medication for IOP, or able to stop such medication for a washout period and the duration of the study without significant risk of adverse consequences related to glaucomatous disease
4. Elevated IOP (≥ 24 and ≤ 34 mm Hg at 8 AM and ≥ 21 and ≤ 34 mm Hg at 10 AM on Screening Two visit and Baseline visit in one or both eyes off treatment

Exclusion Criteria include:

1. Uncontrolled intraocular hypertension defined as >34 mm Hg at either of the screening/baseline visits (after a washout phase in those subjects who were currently receiving ocular hypotensive therapy).
2. Receiving more than one medication for IOP at time of screening.
3. Central corneal thickness of less than 500 µm or greater than 620 µm.
4. BCVA worse than 20/200 in either eye
5. Significant visual field loss (ie, mean deviation > 10 db or field loss within 10 degrees of fixation), a new field defect, or progression of an existing field defect in either eye during the year preceding the study.
6. Acute angle-closure glaucoma or appositional or very narrow anterior chamber angle in either eye.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
intraocular pressure change from baseline. | 4 weeks

SECONDARY OUTCOMES:
Adverse events as a measure of safety/tolerability | 4 weeks
IOP assessments at weekly visits | Weeks 1, 2, 3, 4

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Artesia Clinical Site - Site 02, Artesia, California
  - Inglewood Clinical Site - Site 03, Inglewood, California
  - Petaluma Clinical Site - Site 05, Petaluma, California
  - New Haven Clinical Site - Site 01, New Haven, Connecticut
  - Atlanta Clinical Site - Site 04, Atlanta, Georgia
  - High Point Clinical Site - Site 06, High Point, North Carolina